CLINICAL TRIAL: NCT00413972
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Parallel Groups Study Comparing the Efficacy and Safety of Vytorin Versus Placebo in Subjects With Primary Hypercholesterolemia
Brief Title: Effects of Vytorin Versus Placebo in Subjects With Primary Hypercholesterolemia (Study P04420)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Schering-Plough (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04420; SCH 465981
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Results first posted 2010-05-25 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Vytorin 10/10 (Experimental): Ezetimibe 10 mg with Simvastatin 10 mg
  Interventions: Drug: ezetimibe with simvastatin
- Vytorin 10/20 (Experimental): Ezetimibe 10 mg with Simvastatin 20 mg
  Interventions: Drug: Ezetimibe with Simvastatin
- Vytorin 10/40 (Experimental): Ezetimibe 10 mg with Simvastatin 40 mg
  Interventions: Drug: Ezetimibe with Simvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ezetimibe with simvastatin — Ezetimibe 10 mg with Simvastatin 10 mg once daily for a total of eight weeks
  Arms: Vytorin 10/10
Drug: Ezetimibe with Simvastatin — Ezetimibe 10 mg with Simvastatin 20 mg once daily for a total of eight weeks
  Arms: Vytorin 10/20
Drug: Ezetimibe with Simvastatin — Ezetimibe 10 mg with Simvastatin 40 mg once daily for a total of eight weeks
  Arms: Vytorin 10/40
Drug: Placebo — Placebo once daily for a total of eight weeks
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group Phase 3 study of Vytorin 10/10 (ezetimibe 10 mg with simvastatin 10 mg), Vytorin 10/20 (ezetimibe 10 mg with simvastatin 20 mg), and Vytorin 10/40 (ezetimibe 10 mg with simvastatin 40 mg) compared to placebo administered daily for 8 consecutive weeks in subjects with primary hypercholesterolemia (LDL-C >3.64 mmol/L [140 mg/dL]). The efficacy of daily Vytorin versus placebo in reducing the concentration of LDL-C will be evaluated, and the efficacy of daily Vytorin versus placebo with respect to change in the concentrations of total cholesterol, triglycerides, and HDL-C will be compared. The safety of Vytorin versus placebo will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be >=18 years and <=75 years of age, male or female.
* Primary hypercholesterolemic subject with a plasma LDL cholesterol concentration >3.64 mmol/L (140 mg/dL) to <=6.3 mmol/L (250 mg/dL) using the Friedewald calculation; total cholesterol (TC) >5.2 mmol/L (200 mg/dL) to <12.7 mmol/L (500 mg/dL) and triglyceride concentrations of <=3.99 mmol/L (350 mg/dL) should be met at the same time. At the time of recruitment (Visit 1), these values may be lower if the subject is on lipid-lowering therapy. (ie, prior to the start of lipid lowering drug washout) or may be higher at the start of dietary therapy.
* Liver transaminases (ALT, AST) <=50% above the upper limit of normal, with no active liver disease and CK <=50% above the upper limit of normal.
* Clinical laboratory tests (complete blood count [CBC], blood chemistries, urinalysis) must be within normal limits, or clinically acceptable to the investigator/sponsor.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control.
* Subjects must be free of any clinically significant diseases other than hyperlipidemia that would interfere with study evaluations.
* Subjects must understand and be able to adhere to the dosing and visit schedules.
* Subject must agree to remain on a cholesterol-lowering diet for the duration of the study (according to China Adult Treatment Panel of High Blood Cholesterol).

Exclusion Criteria:

* Subjects whose body mass index (BMI=weight [kg]/height2 [m]) is >=30 kg/m2 at Visit 3 (Baseline Visit).
* Subjects who have known hypersensitivity to HMG CoA reductase inhibitors.
* Subjects who consume >14 alcoholic drinks per week. (A drink is: a can of beer, glass of wine, or single measure of spirits).
* Any condition or situation, which in the opinion of the investigator, might pose a risk to the subject or interfere with participation in the study.
* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.
* Congestive heart failure defined by NYHA as Class III or IV.
* Uncontrolled cardiac arrhythmia.
* Myocardial infarction, coronary bypass surgery, or angioplasty within 6 months of study entry.
* Unstable or severe peripheral artery disease within 3 months of study entry.
* Unstable angina pectoris within 6 months of study entry.
* Uncontrolled hypertension (treated or untreated) with systolic blood pressure >160 mm Hg or diastolic >100 mm Hg at study entry.
* Uncontrolled (as determined by fasting glucose >180 mg/mL or HbA1c >9%) or newly diagnosed (within 1 month of study entry) diabetes mellitus.
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins, ie, secondary causes of hyperlipidemia, such as secondary hypercholesterolemia due to hypothyroidism (thyroid stimulating hormone [TSH] above upper limit of normal). Subjects with a history of hypothyroidism who are on a stable therapy of thyroid hormone replacement for at least 6 weeks are eligible for enrollment if TSH levels are within normal limits before enrollment.
* Known impaired renal function (plasma creatinine >2.0 mg/dL), or nephrotic syndrome at study entry.
* Disorders of the hematologic, digestive, or central nervous systems, including cerebrovascular disease and degenerative disease that would limit study evaluation or participation.
* Known HIV positive.
* Cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas).
* History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Female subject receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vytorin 10/10 | Vytorin 10/20 | Vytorin 10/40 | Placebo
Started | 98 (1 of the 98 randomized subjects was not treated and was excluded from the ITT data set.) | 98 (1 of the 98 randomized subjects was not treated and was excluded from the ITT data set.) | 98 | 98 (1 of the 98 randomized subjects was not treated and was excluded from the ITT data set.)
Completed | 91 | 90 | 88 | 95
Not Completed | 7 | 8 | 10 | 3
Not completed — Adverse Event | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 7 | 2
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vytorin 10/10 | Vytorin 10/20 | Vytorin 10/40 | Placebo | Total
Number analyzed (Participants) | 97 | 97 | 98 | 97 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (10.7) | 57.4 (9.7) | 56.4 (10.3) | 60.2 (9.2) | 58.2 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 61 | 66 | 60 | 246
  Male | 38 | 36 | 32 | 37 | 143
Region of Enrollment [Number; unit: participants]
  China | 97 | 97 | 98 | 97 | 389

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Endpoint After 8 Weeks of Treatment
Time Frame: Baseline, 8 weeks
Population: The number of participants for analysis included those from the ITT data set. 392 subjects were randomized in the study, but 3 of the randomized subjects were not treated and were excluded from the ITT data set. Therefore, only 389 subjects were included in the ITT data set.
Measure: Mean (Standard Error); unit: percent change of LDL-C
Arm/Group | Vytorin 10/10 | Vytorin 10/20 | Vytorin 10/40 | Placebo
Number analyzed (Participants) | 97 | 97 | 98 | 97
percent change of LDL-C | -41.69 (2.06) | -46.83 (2.08) | -49.10 (2.07) | -7.53 (2.04)
Statistical Analysis 1: Comparison: Vytorin 10/10 vs Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: Vytorin 10/20 vs Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: Vytorin 10/40 vs Placebo; Test type: Superiority or Other; p < .0001, ANOVA

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Vytorin 10/10 | Vytorin 10/20 | Vytorin 10/40 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/97 | 0/98 | 0/97
Other Adverse Events (participants affected / at risk) | 0/97 | 0/97 | 0/98 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes